CLINICAL TRIAL: NCT02475109
Title: A Phase 1 Open-Label, Single-Center Study to Evaluate the Safety and Tolerability of Topical Ocular PAN-90806 in Patients With Proliferative Diabetic Retinopathy (PDR)
Brief Title: Study of Topical Ocular PAN-90806 in PDR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PanOptica, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAN-01-201
Record Dates: First submitted 2015-06-13; First posted 2015-06-18 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Diabetic Retinopathy
Keywords: Proliferative Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PAN-90806 Ophthalmic Solution (Experimental): PAN-90806 Ophthalmic Solution taken daily for 8 weeks.
  Interventions: Drug: PAN-90806 Ophthalmic Solution

INTERVENTIONS:
Drug: PAN-90806 Ophthalmic Solution
  Other Names: PAN-90806 Eye Drops

SUMMARY:
The objective of this study is to assess the safety and tolerability of topical ocular PAN-90806 in patients with proliferative diabetic retinopathy.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older with type 1 or type 2 diabetes
* Proliferative diabetic retinopathy (PDR) in study eye retina with or without diabetic macular edema (DME) involving the center of the macula
* Demonstrate the ability, or have a family member who is willing and able, to instill topical ocular drops in the study eye

Exclusion Criteria:

* Current or recent use (within the last 3 months) of anti-vascular endothelial growth factors (anti-VEGF) in either eye;
* Uncontrolled hypertension despite use of antihypertensive medications
* Unwillingness to refrain from wearing contact lenses for the duration of the study.
* Participation in any investigational drug or device study, systemic or ocular, within past 3 months
* Women who are pregnant or nursing
* Known serious allergies or hypersensitivity to the fluorescein dye used in angiography or to the components of the PAN-90806 formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-08; Primary Completion 2016-05 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Adverse Events | 2 months
  Safety will be assessed based upon the incidence of all adverse events, ocular and systemic

SECONDARY OUTCOMES:
The mean change in best-corrected visual acuity from baseline | Week 8
Change in preretinal neovascularization | Week 4 and Week 8
  descriptive observations of the presence and extent as determined by ultra-wide field fluorescein angiography (FA) and color fundus photography (FP)
The mean number of rescue treatments during the study | Week 8
Time to first rescue treatment | up to Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Victor H Gonzalez, M.D., Principal Investigator — Valley Retina Institute
Locations (2):
- United States (2):
  - Valley Retina Institute, Harlingen, Texas
  - Valley Retina Institute, McAllen, Texas

IPD SHARING:
Plan to Share IPD: Undecided